CLINICAL TRIAL: NCT01745237
Title: Detection and Prognostic Significance of Myocardial Damage Visualized by Delayed-Enhancement Cardiovascular Magnetic Resonance in Patients With Sarcoidosis
Brief Title: Delayed-Enhancement Cardiovascular Magnetic Resonance in Patients With Sarcoidosis
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008224; DCMRC-8224a (Other: DUMC)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Cardiac Magnetic Resonance
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study was to determine the ability of cardiac magnetic resonance (CMR) to identify cardiac involvement in patients with sarcoidosis. Patients were to undergo CMR in addition to routine clinical evaluation.

DETAILED DESCRIPTION:
In patients with sarcoidosis, cardiac death is a leading cause of mortality which may represent unrecognized cardiac involvement. Cardiovascular magnetic resonance (CMR) can detect cardiac involvement including minute amounts of myocardial damage. Therefore, the objective of this study was to determine the usefulness of CMR and compare it with standard clinical evaluation for cardiac involvement. Patients with documented extracardiac sarcoidosis or clinically suspected cardiac sarcoidosis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis
* Suspected cardiac sarcoidosis

Exclusion Criteria:

* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven sarcoidosis or suspected cardiac sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 27000 (Estimated)
Dates: Start 2002-09 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
cardiac mortality | > 1year
arrhythmic death | > 1year
Pulmonary mortality | > 1year
  only in subset of patients with pulmonary sarcoidosis

SECONDARY OUTCOMES:
all-cause mortality | > 1year
arrhythmic events | > 1year
Pulmonary Transplant | > 1 year
Cardiac Transplant | > 1 year
PPM placement/high grade AV block | > 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J Kim, MD, Principal Investigator — Duke Cardiovascular Magnetic Resonance Center, Duke University Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Patel MR, Cawley PJ, Heitner JF, Klem I, Parker MA, Jaroudi WA, Meine TJ, White JB, Elliott MD, Kim HW, Judd RM, Kim RJ. Detection of myocardial damage in patients with sarcoidosis. Circulation. 2009 Nov 17;120(20):1969-77. doi: 10.1161/CIRCULATIONAHA.109.851352. Epub 2009 Nov 2. PMID 19884472